CLINICAL TRIAL: NCT01332994
Title: Efficacy and Safety Study of a Sequential Therapy of Tocilizumab (TCZ) and, if Initially Inadequately Responded to Tocilizumab (TCZ), Followed by Rituximab (RTX) in DMARD-IR Patients With Rheumatoid Arthritis (MIRAI)
Brief Title: A Study of RoActemra/Actemra and, if Initially Inadequately Responded to RoActemra/Actemra, Followed by MabThera/Rituxan in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22985
Record Dates: First submitted 2011-03-18; First posted 2011-04-11 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; tocilizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1 g intravenously at Week 16 and 18
  Arms: 2
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously every 4 weeks for 12 weeks.
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously every 4 weeks from Week 16 to Week 28
  Arms: 1

SUMMARY:
This open-label, multi-center, two-arm, uncontrolled and non-randomized study will evaluate the efficacy and safety of RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Patients will receive 8 mg/kg RoActemra/Actemra intravenously every 4 weeks for 12 weeks and - if adequately responded - for further 12 weeks. Patients, who show an inadequate clinical response after the first 12 weeks to RoActemra/Actemra, will receive 1 g MabThera/Rituxan (rituximab) intravenously at Week 16 and 18. The anticipated time of study treatment is 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years of age
* Body weight < /=130kg
* Active rheumatoid arthritis of at least 6 months duration, diagnosed according to the American College of Rheumatology (ACR) criteria of 1987
* Disease Activity Score (DAS28) of >3.2
* Inadequate clinical response to a stable dose of traditional Disease-Modifying Anti-Rheumatic Drugs (DMARD)
* Have received permitted DMARDs, one or more; current DMARD therapy must have been at stable dose for at least 4 weeks prior to baseline

Exclusion Criteria:

* Prior treatment with TNF-inhibitors or other biologic DMARD
* Major surgery (including joint surgery) within eight weeks prior to baseline or planned major surgery within the study duration
* Functional class IV (American College of Rheumatology classification)
* Rheumatic autoimmune disease other than rheumatoid arthritis
* History of or current inflammatory joint disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- Germany (61):
  - Aachen
  - Bad Aibling
  - Bad Bramstedt
  - Bad Nauheim
  - Bad Staffelstein
  - Bayreuth
  - Berlin
  - Blaubeuren Abbey
  - Bonn
  - Bruchhausen-Vilsen
  - Chemnitz
  - Cologne
  - Donaueschingen
  - Dresden
  - Düsseldorf
  - Erfurt
  - Essen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Giessen
  - Gommern
  - Goslar
  - Göttingen
  - Greifswald
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Hildesheim
  - Hofheim
  - Jena
  - Kiel
  - Leipzig
  - Lingen
  - Ludwigsfelde
  - Mainz
  - Mönchengladbach
  - München
  - Naumburg
  - Naunhof
  - Neuss
  - Nienburg
  - Olsberg
  - Osnabrück
  - Plochingen
  - Potsdam
  - Ratingen
  - Regensburg
  - Rendsburg
  - Rheine
  - Rostock
  - Saarbrücken
  - Sendenhorst
  - Stuttgart
  - Traunstein
  - Trier
  - Tübingen
  - Ulm
  - Wiesbaden
  - Würzburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a screening period of up to 4 weeks, eligible participants were treated according to a predefined treatment algorithm based on disease response. In certain cases a re-screening was allowed. Participants were enrolled into the study with the administration of their first dose.
Groups:
- Tocilizumab (TCZ)/TCZ or TCZ/Rituximab (RTX): All participants were assigned to receive TCZ 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion every 4 weeks for a total of 4 infusions from Baseline to Week 12. Clinical response was assessed at Week 16 using Disease Activity Score Based on 28-Joint Count (DAS28) to determine subsequent treatment assignment. Participants who achieved early remission, defined as a DAS28 score of less than (<) 2.6, were transferred to clinical routine care and no longer received study medication. Participants who were considered partial responders, defined as a decrease from Baseline in DAS28 score greater than (>) 1.2 or a score between 2.6 and 3.2, inclusive, received TCZ 8 mg/kg via IV infusion every 4 weeks for a total of 4 additional infusions from Week 16 to 28. Those with assessed as having no response, defined as a decrease from Baseline in DAS28 score less than or equal to (≤) 1.2 or a score >3.2, received RTX 1000 milligrams (mg) via IV infusion at Weeks 16 and 18.
Period: Overall Study
Arm/Group | Tocilizumab (TCZ)/TCZ or TCZ/Rituximab (RTX)
Started | 519
Completed Week 16 | 463
Completed Week 32 (TCZ/TCZ) | 200
Completed Week 32 (TCZ/RTX) | 26
Completed Week 66 (TCZ/RTX) | 25
Completed | 448
Not Completed | 71
Not completed — Adverse Event | 34
Not completed — Death | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 15
Not completed — Administrative Problem | 2
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Population: Main Intent-to-Treat (ITT) Population: All participants who received at least one dose of TCZ.
Groups:
- TCZ/TCZ or TCZ/RTX: All participants were assigned to receive TCZ 8 mg/kg via IV infusion every 4 weeks for a total of 4 infusions from Baseline to Week 12. Clinical response was assessed at Week 16 using DAS28 to determine subsequent treatment assignment. Participants who achieved early remission, defined as a DAS28 score of <2.6, were transferred to clinical routine care and no longer received study medication. Participants who were considered partial responders, defined as a decrease from Baseline in DAS28 score >1.2 or a score between 2.6 and 3.2, inclusive, received TCZ 8 mg/kg via IV infusion every 4 weeks for a total of 4 additional infusions from Week 16 to 28. Those with assessed as having no response, defined as a decrease from Baseline in DAS28 score ≤1.2 or a score >3.2, received RTX 1000 mg via IV infusion at Weeks 16 and 18.
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352
  Male | 167

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Remission at Week 16 According to DAS28
Description: The DAS28 was calculated as [0.28 times (x) the square root of number of swollen joints] plus (+) [0.56 x the square root of number of tender joints] + [0.7 x the natural log of erythrocyte sedimentation rate (ESR)] + [0.014 x Visual Analog Scale (VAS) patient global assessment of disease activity]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' DAS28 scores ranged from 0 to 10, with higher scores indicating increased disease activity. Remission was defined as a DAS28 score <2.6 at the assessment visit.
Time Frame: Week 16
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants | 42.8 [38.5 to 47.2]
Statistical Analysis 1: Comparison: TCZ/TCZ or TCZ/RTX; Test type: Superiority or Other; p = 0.1648, Exact one-sided binomial test — Exact one-sided binomial test on single proportions with a significance level of alpha equals (=) 0.025. Null hypothesis: Proportion of participants reaching DAS28 remission (<2.6) at Week 16 is ≤45 percent (%)

2. Secondary Outcome: Percentage of Participants Achieving Remission According to DAS28 at Weeks 4, 8, and 12
Description: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x VAS patient global assessment of disease activity]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' DAS28 scores ranged from 0 to 10, with higher scores indicating increased disease activity. Remission was defined as a DAS28 score <2.6 at the assessment visit.
Time Frame: Weeks 4, 8, and 12
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants
  Week 4 | 21.6 [18.1 to 25.4]
  Week 8 | 40.1 [35.8 to 44.4]
  Week 12 | 43.2 [38.9 to 47.5]

3. Secondary Outcome: Percentage of Participants Achieving Remission According to DAS28 at Weeks 16, 20, 24, and 28 Among Participants Treated With 8 Courses of Tocilizumab
Description: as for outcome 2
Time Frame: Weeks 16, 20, 24, and 28
Population: ITT2 Population: All participants who received at least one dose of TCZ in the first treatment period with at least one efficacy measurement under TCZ, receiving TCZ in the second treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 213
percentage of participants
  Week 16 | 1.4 [0.3 to 4.1]
  Week 20 | 41.3 [34.6 to 48.2]
  Week 24 | 51.2 [44.3 to 58.1]
  Week 28 | 55.9 [48.9 to 62.6]

4. Secondary Outcome: Percentage of Participants Achieving Remission According to DAS28 at Week 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: as for outcome 2
Time Frame: Week 32
Population: ITT2 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 213
percentage of participants | 54.9 [48.0 to 61.7]

5. Secondary Outcome: Percentage of Participants Achieving Remission According to DAS28 at Week 32 Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 2
Time Frame: Week 32
Population: ITT3 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
percentage of participants | 14.8 [4.2 to 33.7]

6. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity Score (LDAS) According to DAS28
Description: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x the patient global assessment of disease activity using a VAS]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' DAS28 scores ranged from 0 to 10, with higher scores indicating increased disease activity. LDAS was defined as a DAS28 score <3.2 at the assessment visit.
Time Frame: Week 16
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants | 68.8 [64.6 to 72.8]

7. Secondary Outcome: Percentage of Participants Achieving LDAS According to DAS28 Among Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 6
Time Frame: Week 32
Population: ITT3 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
percentage of participants | 33.3 [16.5 to 54.0]

8. Secondary Outcome: Percentage of Participants Achieving a Clinically Relevant Reduction From Baseline in DAS28 at Week 16
Description: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x VAS patient global assessment of disease activity]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' DAS28 scores ranged from 0 to 10, with higher scores indicating increased disease activity. Reductions >1.2 points from Baseline to the assessment visit were considered clinically relevant.
Time Frame: Baseline and Week 16
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants | 86.1 [82.9 to 89.0]

9. Secondary Outcome: Percentage of Participants Achieving a Clinically Relevant Reduction From Baseline in DAS28 at Weeks 4, 8, and 12
Description: as for outcome 8
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants
  Week 4 | 74.6 [70.6 to 78.3]
  Week 8 | 81.5 [77.9 to 84.8]
  Week 12 | 83.4 [79.9 to 86.5]

10. Secondary Outcome: Percentage of Participants Achieving a Clinically Relevant Reduction in DAS28 From Week 16 to Week 32 Among Nonresponding Participants Treated With Rituximab
Description: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x VAS patient global assessment of disease activity]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' DAS28 scores ranged from 0 to 10, with higher scores indicating increased disease activity. Reductions >1.2 points from the reference visit (Week 16) to the assessment visit were considered clinically relevant.
Time Frame: Weeks 16 and 32
Population: ITT3 Population: All participants who received at least one dose of TCZ in the first treatment period and at least one dose of RTX in the second treatment period with at least one efficacy measurement under RTX.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
percentage of participants | 37.0 [19.4 to 57.6]

11. Secondary Outcome: DAS28 Scores During and After Treatment
Description: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x VAS patient global assessment of disease activity]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' DAS28 scores ranged from 0 to 10, with higher scores indicating increased disease activity.
Time Frame: Baseline and Weeks 4, 8, 12, 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 516
units on a scale
  Baseline (n=516) | 5.7 (1.0)
  Week 4 (n=508) | 3.6 (1.3)
  Week 8 (n=491) | 3.0 (1.4)
  Week 12 (n=483) | 2.8 (1.4)
  Week 16 (n=485) | 2.6 (1.3)

12. Secondary Outcome: DAS28 Scores During and After Treatment Among Participants Treated With 8 Courses of Tocilizumab
Description: as for outcome 11
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 213
units on a scale
  Baseline (n=213) | 6.0 (0.9)
  Week 4 (n=213) | 4.0 (1.2)
  Week 8 (n=205) | 3.4 (1.2)
  Week 12 (n=207) | 3.3 (1.1)
  Week 16 (n=213) | 3.3 (0.6)
  Week 20 (n=206) | 2.8 (1.0)
  Week 24 (n=197) | 2.6 (1.1)
  Week 28 (n=200) | 2.4 (1.1)
  Week 32 (n=193) | 2.5 (1.2)

13. Secondary Outcome: DAS28 Scores During and After Treatment Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 11
Time Frame: Baseline and Weeks 4, 8, 12, 16, 24, and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
units on a scale
  Baseline (n=27) | 5.7 (1.0)
  Week 4 (n=27) | 4.5 (1.2)
  Week 8 (n=26) | 4.2 (1.5)
  Week 12 (n=27) | 4.8 (1.6)
  Week 16 (n=27) | 5.1 (1.2)
  Week 24 (n=26) | 4.6 (1.4)
  Week 32 (n=26) | 4.0 (1.5)

14. Secondary Outcome: DAS28 Scores During Safety Follow-Up Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 11
Time Frame: Weeks 40, 48, 56, and 66
Population: ITT3 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 26
units on a scale
  Week 40 (n=26) | 3.9 (1.5)
  Week 48 (n=25) | 3.9 (1.2)
  Week 56 (n=22) | 4.1 (1.8)
  Week 66 (n=25) | 3.9 (1.5)

15. Secondary Outcome: Percentage of Participants Achieving a Response According to European League Against Rheumatism (EULAR) Criteria at Weeks 4, 8, 12 and 16
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the assessment visit and the DAS28 reduction from Baseline. Participants with a score ≤3.2 and reduction of >1.2 points were assessed as having a 'good' response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a 'moderate' response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as nonresponders with response recorded as 'none.'
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants
  Week 4, Good | 36.0 [31.9 to 40.3]
  Week 4, Moderate | 47.8 [43.4 to 52.2]
  Week 4, None | 16.2 [13.1 to 19.6]
  Week 8, Good | 56.1 [51.7 to 60.4]
  Week 8, Moderate | 30.6 [26.7 to 34.8]
  Week 8, None | 13.3 [10.5 to 16.5]
  Week 12, Good | 61.1 [56.7 to 65.3]
  Week 12, Moderate | 25.6 [21.9 to 29.6]
  Week 12, None | 13.3 [10.5 to 16.5]
  Week 16, Good | 68.2 [64.0 to 72.2]
  Week 16, Moderate | 20.2 [16.9 to 23.9]
  Week 16, None | 11.6 [8.9 to 14.6]

16. Secondary Outcome: Percentage of Participants Achieving a Response According to EULAR Criteria at Week 32 Compared to Week 16 Among Nonresponding Participants Treated With Rituximab
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the assessment visit and the DAS28 reduction from the reference visit (Week 16). Participants with a score ≤3.2 and reduction of >1.2 points were assessed as having a 'good' response. Participants with a score >3.2 with reduction of >1.2 points, or a score ≤5.1 with reduction of >0.6 to ≤1.2 points, were assessed as having a 'moderate' response. Participants with a score >5.1 with reduction of >0.6 to ≤1.2 points, or any score with reduction ≤0.6 points, were assessed as nonresponders with response recorded as 'none.'
Time Frame: Weeks 16 and 32
Population: ITT3 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
percentage of participants
  Good | 25.9 [11.1 to 46.3]
  Moderate | 29.6 [13.8 to 50.2]
  None | 44.4 [25.5 to 64.7]

17. Secondary Outcome: Percentage of Participants Achieving a Response According to EULAR Criteria at Weeks 20, 24, 28, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: as for outcome 15
Time Frame: Baseline and Weeks 20, 24, 28, and 32
Population: ITT2 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 213
percentage of participants
  Week 20, Good | 65.3 [58.5 to 71.6]
  Week 20, Moderate | 30.0 [24.0 to 36.7]
  Week 20, None | 4.7 [2.3 to 8.5]
  Week 24, Good | 68.1 [61.4 to 74.3]
  Week 24, Moderate | 23.9 [18.4 to 30.3]
  Week 24, None | 8.0 [4.7 to 12.5]
  Week 28, Good | 72.8 [66.3 to 78.6]
  Week 28, Moderate | 19.2 [14.2 to 25.2]
  Week 28, None | 8.0 [4.7 to 12.5]
  Week 32, Good | 66.7 [59.9 to 73.0]
  Week 32, Moderate | 20.7 [15.4 to 26.7]
  Week 32, None | 12.7 [8.5 to 17.9]

18. Secondary Outcome: Percentage of Participants Achieving a Response According to American College of Rheumatology (ACR) Criteria at Weeks 4, 8, 12, and 16
Description: Response was determined using ACR criteria based upon assessment of 66 joints for swelling and 68 joints for tenderness; joints were classified dichotomously as swollen or not swollen and tender or not tender. Respectively, these assessments were used to generate a swollen joint count (SJC) ranging from 0 to 66 swollen joints and a tender joint count (TJC) ranging from 0 to 68 tender joints. Response was defined as a reduction from Baseline of at least 20% for one of the following: VAS scores for patient-reported pain, patient global assessment of disease activity, or physician global assessment of disease activity, Health Assessment Questionnaire Disability Index (HAQ-DI), or C-reactive protein (CRP); plus a reduction in individual SJC and TJC of 20% (ACR20), 50% (ACR50), or 70% (ACR70). VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.'
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Main ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants
  Week 4, ACR20 | 39.1 [34.9 to 43.5]
  Week 4, ACR50 | 15.0 [12.1 to 18.4]
  Week 4, ACR70 | 5.8 [3.9 to 8.1]
  Week 8, ACR20 | 61.1 [56.7 to 65.3]
  Week 8, ACR50 | 33.5 [29.5 to 37.8]
  Week 8, ACR70 | 15.2 [12.2 to 18.6]
  Week 12, ACR20 | 64.0 [59.7 to 68.1]
  Week 12, ACR50 | 42.8 [38.5 to 47.2]
  Week 12, ACR70 | 20.2 [16.9 to 23.9]
  Week 16, ACR20 | 67.1 [62.8 to 71.1]
  Week 16, ACR50 | 45.7 [41.3 to 50.1]
  Week 16, ACR70 | 24.5 [20.8 to 28.4]

19. Secondary Outcome: Percentage of Participants Achieving a Response According to ACR Criteria at Week 32 Compared to Week 16 Among Nonresponding Participants Treated With Rituximab
Description: Response was determined using ACR criteria based upon assessment of 66 joints for swelling and 68 joints for tenderness; joints were classified dichotomously as swollen or not swollen and tender or not tender. Respectively, these assessments were used to generate an SJC ranging from 0 to 66 swollen joints and a TJC ranging from 0 to 68 tender joints. Response was defined as a reduction from the reference visit (Week 16) of at least 20% for one of the following: VAS scores for patient-reported pain, patient global assessment of disease activity, or physician global assessment of disease activity, HAQ-DI, or CRP; plus a reduction in individual SJC and TJC of 20% (ACR20), 50% (ACR50), or 70% (ACR70). VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.'
Time Frame: Weeks 16 and 32
Population: ITT3 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
percentage of participants
  ACR20 | 40.7 [22.4 to 61.2]
  ACR50 | 33.3 [16.5 to 54.0]
  ACR70 | 22.2 [8.6 to 42.3]

20. Secondary Outcome: Percentage of Participants Achieving a Response According to ACR Criteria at Weeks 20, 24, 28, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: Response was determined using ACR criteria based upon assessment of 66 joints for swelling and 68 joints for tenderness; joints were classified dichotomously as swollen or not swollen and tender or not tender. Respectively, these assessments were used to generate an SJC ranging from 0 to 66 swollen joints and a TJC ranging from 0 to 68 tender joints. Response was defined as a reduction from Baseline of at least 20% for one of the following: VAS scores for patient-reported pain, patient global assessment of disease activity, or physician global assessment of disease activity, HAQ-DI, or CRP; plus a reduction in individual SJC and TJC of 20% (ACR20), 50% (ACR50), or 70% (ACR70). VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.'
Time Frame: Baseline and Weeks 20, 24, 28, and 32
Population: ITT2 Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 213
percentage of participants
  Week 20, ACR20 | 74.2 [67.8 to 79.9]
  Week 20, ACR50 | 45.1 [38.3 to 52.0]
  Week 20, ACR70 | 21.1 [15.8 to 27.2]
  Week 24, ACR20 | 72.8 [66.3 to 78.6]
  Week 24, ACR50 | 49.8 [42.9 to 56.7]
  Week 24, ACR70 | 21.6 [16.3 to 27.7]
  Week 28, ACR20 | 73.2 [66.8 to 79.1]
  Week 28, ACR50 | 53.1 [46.1 to 59.9]
  Week 28, ACR70 | 30.5 [24.4 to 37.2]
  Week 32, ACR20 | 75.6 [69.2 to 81.2]
  Week 32, ACR50 | 54.9 [48.0 to 61.7]
  Week 32, ACR70 | 34.3 [27.9 to 41.1]

21. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) and Simplified Disease Activity Index (SDAI) Scores at Weeks 4, 8, 12, and 16
Description: The CDAI was calculated as [SJC + TJC + VAS patient global assessment of disease activity + VAS physician global assessment of disease activity]. VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity.' CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity. The SDAI was determined by adding CRP level to the CDAI score. Scores ranged from 0 to 86, with higher scores also indicating increased disease activity. A reduction in either score at the assessment visit reflects improvement in disease.
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 509
units on a scale
  CDAI, Week 4 (n=509) | -10.9 (10.2)
  CDAI, Week 8 (n=497) | -16.5 (11.1)
  CDAI, Week 12 (n=486) | -18.3 (11.5)
  CDAI, Week 16 (n=485) | -19.4 (11.5)
  SDAI, Week 4 (n=496) | -12.3 (10.6)
  SDAI, Week 8 (n=489) | -17.9 (11.5)
  SDAI, Week 12 (n=474) | -19.7 (11.9)
  SDAI, Week 16 (n=471) | -20.7 (12.2)

22. Secondary Outcome: Change From Week 16 to 32 in CDAI and SDAI Scores Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 21
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 25
units on a scale
  CDAI (n=25) | -14.2 (12.0)
  SDAI (n=24) | -14.0 (12.5)

23. Secondary Outcome: Change From Baseline in CDAI and SDAI Scores at Weeks 20, 24, 28, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: as for outcome 21
Time Frame: Baseline and Weeks 20, 24, 28, and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 208
units on a scale
  CDAI, Week 20 (n=208) | -21.7 (11.7)
  CDAI, Week 24 (n=199) | -22.8 (11.4)
  CDAI, Week 28 (n=200) | -24.6 (12.5)
  CDAI, Week 32 (n=194) | -24.0 (13.4)
  SDAI, Week 20 (n=200) | -22.9 (12.5)
  SDAI, Week 24 (n=190) | -24.3 (12.1)
  SDAI, Week 28 (n=195) | -25.9 (13.2)
  SDAI, Week 32 (n=189) | -25.2 (14.0)

24. Secondary Outcome: Change From Baseline in Hemoglobin at Weeks 4, 8, 12, and 16
Description: Blood samples for laboratory assessments, including hemoglobin level, were collected prior to each dose of study medication. The mean hemoglobin level was determined at Baseline and for assessment visits by averaging the observed hemoglobin level among all participants providing evaluable blood samples. Change from Baseline was calculated as [mean hemoglobin at the assessment visit minus mean hemoglobin at Baseline] and expressed in grams per liter (g/L).
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 509
g/L
  Week 4 (n=509) | 4.9 (7.2)
  Week 8 (n=496) | 6.4 (8.8)
  Week 12 (n=483) | 6.9 (9.1)
  Week 16 (n=477) | 7.5 (9.1)

25. Secondary Outcome: Change From Baseline in CRP at Weeks 4, 8, 12, and 16
Description: Blood samples for laboratory assessments, including CRP level, were collected prior to each dose of study medication. The mean CRP level was determined at Baseline and for assessment visits by averaging the observed CRP level among all participants providing evaluable blood samples. Change from Baseline was calculated as [mean CRP at the assessment visit minus mean CRP at Baseline] and expressed in milligrams per deciliter (mg/dL).
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 497
mg/dL
  Week 4 (n=497) | -1.4 (1.9)
  Week 8 (n=492) | -1.4 (1.9)
  Week 12 (n=476) | -1.4 (1.9)
  Week 16 (n=471) | -1.3 (1.9)

26. Secondary Outcome: Change From Baseline in ESR at Weeks 4, 8, 12, and 16
Description: Blood samples for laboratory assessments, including ESR, were collected prior to each dose of study medication. The mean ESR was determined at Baseline and for assessment visits by averaging the observed ESR among all participants providing evaluable blood samples. Change from Baseline was calculated as [mean ESR at the assessment visit minus mean ESR at Baseline] and expressed in millimeters per hour (mm/h).
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 507
mm/h
  Week 4 (n=507) | -25.2 (18.1)
  Week 8 (n=494) | -26.6 (18.9)
  Week 12 (n=484) | -26.3 (19.1)
  Week 16 (n=484) | -27.5 (18.7)

27. Secondary Outcome: Change in Hemoglobin From Week 16 to 32 Among Nonresponding Participants Treated With Rituximab
Description: Blood samples for laboratory assessments, including hemoglobin level, were collected prior to each dose of study medication. The mean hemoglobin level was determined at Baseline and for assessment visits by averaging the observed hemoglobin level among all participants providing evaluable blood samples. Change was calculated as [mean hemoglobin at Week 32 minus mean hemoglobin at Week 16] and expressed in g/L.
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 26
g/L | -2.0 (8.3)

28. Secondary Outcome: Change in CRP From Week 16 to 32 Among Nonresponding Participants Treated With Rituximab
Description: Blood samples for laboratory assessments, including CRP level, were collected prior to each dose of study medication. The mean CRP level was determined at Baseline and for assessment visits by averaging the observed CRP level among all participants providing evaluable blood samples. Change was calculated as [mean CRP at Week 32 minus mean CRP at Week 16] and expressed in mg/dL.
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 25
mg/dL | 0.7 (1.7)

29. Secondary Outcome: Change in ESR From Week 16 to 32 Among Nonresponding Participants Treated With Rituximab
Description: Blood samples for laboratory assessments, including ESR, were collected prior to each dose of study medication. The mean ESR was determined at Baseline and for assessment visits by averaging the observed ESR among all participants providing evaluable blood samples. Change was calculated as [mean ESR at Week 32 minus mean ESR at Week 16] and expressed in mm/h.
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 26
mm/h | 11.5 (17.9)

30. Secondary Outcome: Change From Baseline in Hemoglobin at Weeks 20, 24, 28, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: Blood samples for laboratory assessments, including hemoglobin level, were collected prior to each dose of study medication. The mean hemoglobin level was determined at Baseline and for assessment visits by averaging the observed hemoglobin level among all participants providing evaluable blood samples. Change from Baseline was calculated as [mean hemoglobin at the assessment visit minus mean hemoglobin at Baseline] and expressed in g/L.
Time Frame: Baseline and Weeks 20, 24, 28, and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 207
g/L
  Week 20 (n=207) | 5.5 (9.0)
  Week 24 (n=198) | 6.6 (9.4)
  Week 28 (n=197) | 6.9 (9.5)
  Week 32 (n=197) | 8.3 (10.4)

31. Secondary Outcome: Change From Baseline in CRP at Weeks 20, 24, 28, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: Blood samples for laboratory assessments, including CRP level, were collected prior to each dose of study medication. The mean CRP level was determined at Baseline and for assessment visits by averaging the observed CRP level among all participants providing evaluable blood samples. Change from Baseline was calculated as [mean CRP at the assessment visit minus mean CRP at Baseline] and expressed in mg/dL.
Time Frame: Baseline and Weeks 20, 24, 28, and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 200
mg/dL
  Week 20 (n=200) | -1.3 (1.9)
  Week 24 (n=191) | -1.4 (1.9)
  Week 28 (n=195) | -1.3 (1.9)
  Week 32 (n=192) | -1.3 (1.9)

32. Secondary Outcome: Change From Baseline in ESR at Weeks 20, 24, 28, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: Blood samples for laboratory assessments, including ESR, were collected prior to each dose of study medication. The mean ESR was determined at Baseline and for assessment visits by averaging the observed ESR among all participants providing evaluable blood samples. Change from Baseline was calculated as [mean ESR at the assessment visit minus mean ESR at Baseline] and expressed in mm/h.
Time Frame: Baseline and Weeks 20, 24, 28, and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 206
mm/h
  Week 20 (n=206) | -28.6 (17.6)
  Week 24 (n=197) | -29.4 (18.0)
  Week 28 (n=200) | -29.4 (18.1)
  Week 32 (n=196) | -28.6 (20.2)

33. Secondary Outcome: Percentage of Participants Withdrawing From the Study for Insufficient Therapeutic Response
Description: Study discontinuation was documented by reason for each participant prematurely withdrawing from the study. The percentage of participants was calculated as the number withdrawing for insufficient therapeutic response divided by the total number of participants who began treatment.
Time Frame: Baseline to Week 16
Population: Main ITT Population. Participants who withdrew for reasons other than insufficient therapeutic response were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 485
percentage of participants | 0.2 [0.0 to 1.1]

34. Secondary Outcome: Percentage of B-Cells at Baseline by B-Cell Subpopulation Among Participants With Early Remission
Description: Blood samples were collected to analyze total B-cell panel via immunophenotyping. Subpopulations were as follows: transitional (cluster of differentiation [CD] 19-positive, immunoglobulin (Ig) D-positive, CD38 medium, CD10-positive); naive (CD19-positive, IgD-positive, CD38 medium, CD27-negative); pre-switch memory (CD19-positive, CD27-positive, IgD-positive); post-switch memory (CD19-positive, CD27-positive, IgD-negative); IgG-positive class-switched (CD19-positive, IgG-positive); IgA-positive class-switched (CD19-positive, IgA-positive); double-negative memory (CD19-positive, IgD-negative, CD27-negative); and plasmablasts (CD19-positive, IgD-negative, CD38 high, CD27 high). Naive B-cell compartment was defined as the sum of transitional and naive B-cells. The sum of memory B-cell subsets with or without double-negative B-cells was also determined.
Time Frame: Baseline
Population: ITT1 Population: All participants who received at least one dose of TCZ in the first treatment period and who completed the study reaching remission at Week 16. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Median (Full Range); unit: percentage of B-cells
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 196
percentage of B-cells
  Naive B-cell compartment (n=196) | 61.1 [5.3 to 102.9]
  Transitional B-cells (n=196) | 1.4 [0.1 to 18.8]
  Naive B-cells (n=196) | 58.1 [3.4 to 94.2]
  Memory including double-negative (n=46) | 56.4 [20.2 to 103.5]
  Memory excluding double-negative (n=194) | 46.5 [5.6 to 125.8]
  Pre-switch memory B-cells (n=196) | 11.1 [1.3 to 73.6]
  Post-switch memory B-cells (n=196) | 16.4 [0.8 to 58.1]
  IgG-positive class-switched B-cells (n=195) | 9.9 [0.3 to 42]
  IgA-positive class-switched B-cells (n=194) | 7.4 [0.7 to 35.6]
  Double-negative B-cells (n=46) | 6.1 [2.5 to 16.3]
  Plasmablasts (n=196) | 0.3 [0 to 19.9]

35. Secondary Outcome: Percentage of B-Cells at Baseline by B-Cell Subpopulation Among Participants Treated With 8 Courses of Tocilizumab
Description: as for outcome 34
Time Frame: Baseline
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Median (Full Range); unit: percentage of B-cells
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 197
percentage of B-cells
  Naive B-cell compartment (n=197) | 57.1 [5.6 to 91.2]
  Transitional B-cells (n=197) | 1.3 [0.0 to 13.4]
  Naive B-cells (n=197) | 55.5 [4.7 to 87.1]
  Memory including double-negative (n=57) | 63.2 [18.8 to 113.7]
  Memory excluding double-negative (n=196) | 49.7 [10.9 to 120.1]
  Pre-switch memory B-cells (n=197) | 11.6 [0.9 to 74.1]
  Post-switch memory B-cells (n=197) | 17.2 [2.8 to 52.7]
  IgG-positive class-switched B-cells (n=196) | 10 [0.2 to 38.4]
  IgA-positive class-switched B-cells (n=196) | 8.0 [1.4 to 34.4]
  Double-negative B-cells (n=57) | 6.6 [1.2 to 19.1]
  Plasmablasts (n=197) | 0.3 [0 to 7.6]

36. Secondary Outcome: Percentage of B-Cells at Baseline by B-Cell Subpopulation Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 34
Time Frame: Baseline
Population: ITT3 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Median (Full Range); unit: percentage of B-cells
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 25
percentage of B-cells
  Naive B-cell compartment (n=25) | 65.9 [9.8 to 85.0]
  Transitional B-cells (n=25) | 1.6 [0.2 to 7.0]
  Naive B-cells (n=25) | 61.9 [5.8 to 83.4]
  Memory including double-negative (n=4) | 45.1 [37.1 to 86.7]
  Memory excluding double-negative (n=25) | 41.5 [21.6 to 139.6]
  Pre-switch memory B-cells (n=25) | 9.1 [2.4 to 36.2]
  Post-switch memory B-cells (n=25) | 16.1 [6.9 to 64.1]
  IgG-positive class-switched B-cells (n=25) | 8.7 [5.0 to 32.7]
  IgA-positive class-switched B-cells (n=25) | 7.7 [3.4 to 29.3]
  Double-negative B-cells (n=4) | 7.5 [5.9 to 9.1]
  Plasmablasts (n=25) | 0.3 [0.0 to 3.2]

37. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Percentage of B-Cells at Baseline and Difference in DAS28 Scores Between Baseline and Week 16 Among Participants With Early Remission
Description: Blood samples were collected to analyze total B-cell panel via immunophenotyping. Subpopulations were as follows: transitional, naïve, pre-switch memory, post-switch memory, IgG-positive class-switched, IgA-positive class-switched, double-negative memory, and plasmablasts. Naive B-cell compartment was defined as the sum of transitional and naive B-cells. The sum of memory B-cell subsets with or without double-negative B-cells was also determined. Extent of disease response, using change from Baseline to Week 16 in DAS28 score, was correlated to the percentage of B-cells within each subpopulation at Baseline. Correlation is indicated by a correlation coefficient (r) >0.2, with greater values indicating a stronger correlation.
Time Frame: Baseline and Week 16
Population: ITT1 Population; n = number of data pairs included in the analysis.
Measure: Number; unit: coefficient
Units Other Than Participants: Pairs
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 217
Number analyzed (Pairs) | 192
coefficient
  Naive B-cell compartment (n=192) | -0.02258
  Transitional B-cells (n=192) | -0.00949
  Naive B-cells (n=192) | -0.01920
  Memory B-cells (n=62) | -0.03148
  Pre-switch memory B-cells (n=192) | 0.03221
  Post-switch memory B-cells (n=192) | 0.05419
  IgG-positive class-switched B-cells (n=192) | 0.08864
  IgA-positive class-switched B-cells (n=192) | 0.01041
  Double-negative B-cells (n=62) | -0.02134
  Plasmablasts (n=192) | 0.00397
Statistical Analysis 1: Comparison: TCZ/TCZ or TCZ/RTX; Naive B-cell compartment; Test type: Superiority or Other; p = 0.7559, Spearman Rank-Order Correlation; Probability values for the Spearman correlation were calculated as [square root of (n minus 2) x [square root of (r^2 divided by 1 minus r^2)]
Statistical Analysis 2: Comparison: TCZ/TCZ or TCZ/RTX; Transitional B-cells; Test type: Superiority or Other; p = 0.8961, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: TCZ/TCZ or TCZ/RTX; Naive B-cells; Test type: Superiority or Other; p = 0.7915, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 4: Comparison: TCZ/TCZ or TCZ/RTX; Memory B-cells; Test type: Superiority or Other; p = 0.8081, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 5: Comparison: TCZ/TCZ or TCZ/RTX; Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.6574, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 6: Comparison: TCZ/TCZ or TCZ/RTX; Post-switch memory B-cells; Test type: Superiority or Other; p = 0.4553, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 7: Comparison: TCZ/TCZ or TCZ/RTX; IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.2215, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 8: Comparison: TCZ/TCZ or TCZ/RTX; IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.8860, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 9: Comparison: TCZ/TCZ or TCZ/RTX; Double-negative B-cells; Test type: Superiority or Other; p = 0.8693, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 10: Comparison: TCZ/TCZ or TCZ/RTX; Plasmablasts; Test type: Superiority or Other; p = 0.9564, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]

38. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Percentage of B-Cells at Baseline and Difference in DAS28 Scores Between Baseline and Weeks 16, 24, and 32 Among Participants Treated With 8 Courses of Tocilizumab
Description: Blood samples were collected to analyze total B-cell panel via immunophenotyping. Subpopulations were as follows: transitional, naïve, pre-switch memory, post-switch memory, IgG-positive class-switched, IgA-positive class-switched, double-negative memory, and plasmablasts. Naive B-cell compartment was defined as the sum of transitional and naive B-cells. The sum of memory B-cell subsets with or without double-negative B-cells was also determined. Extent of disease response, using change from Baseline in DAS28 score, was correlated to the percentage of B-cells within each subpopulation at Baseline. Correlation is indicated by a correlation coefficient (r) >0.2, with greater values indicating a stronger correlation.
Time Frame: Baseline and Weeks 16, 24, and 32
Population: ITT2 Population; n = number of data pairs included in the analysis.
Measure: Number; unit: coefficient
Units Other Than Participants: Pairs
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 213
Number analyzed (Pairs) | 199
coefficient
  Week 16, Naive B-cell compartment (n=199) | 0.00007
  Week 16, Transitional B-cells (n=199) | -0.06529
  Week 16, Naive B-cells (n=199) | 0.02334
  Week 16, Memory B-cells (n=75) | 0.03478
  Week 16, Pre-switch memory B-cells (n=199) | -0.01889
  Week 16, Post-switch memory B-cells (n=199) | -0.04161
  Week 16, IgG-positive class-switched (n=199) | -0.06235
  Week 16, IgA-positive class-switched (n=199) | -0.06492
  Week 16, Double-negative B-cells (n=75) | -0.04352
  Week 16, Plasmablasts (n=199) | -0.13161
  Week 24, Naive B-cell compartment (n=162) | -0.18469
  Week 24, Transitional B-cells (n=162) | -0.21966
  Week 24, Naive B-cells (n=162) | -0.15683
  Week 24, Memory B-cells (n=76) | 0.15135
  Week 24, Pre-switch memory B-cells (n=162) | 0.08074
  Week 24, Post-switch memory B-cells (n=162) | 0.10798
  Week 24, IgG-positive class-switched (n=161) | 0.10752
  Week 24, IgA-positive class-switched (n=162) | 0.11023
  Week 24, Double-negative B-cells (n=76) | 0.05609
  Week 24, Plasmablasts (n=162) | 0.07468
  Week 32, Naive B-cell compartment (n=179) | -0.12635
  Week 32, Transitional B-cells (n=179) | -0.09234
  Week 32, Naive B-cells (n=179) | -0.11114
  Week 32, Memory B-cells (n=88) | 0.05361
  Week 32, Pre-switch memory B-cells (n=179) | 0.12265
  Week 32, Post-switch memory B-cells (n=179) | 0.05867
  Week 32, IgG-positive class-switched (n=181) | 0.06381
  Week 32, IgA-positive class-switched (n=181) | 0.06036
  Week 32, Double-negative B-cells (n=90) | -0.06310
  Week 32, Plasmablasts (n=179) | 0.02205
Statistical Analysis 1: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Naive B-cell compartment; Test type: Superiority or Other; p = 0.9993, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 2: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Transitional B-cells; Test type: Superiority or Other; p = 0.3596, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Naive B-cells; Test type: Superiority or Other; p = 0.7435, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 4: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Memory B-cells; Test type: Superiority or Other; p = 0.7671, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 5: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.7912, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 6: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Post-switch memory B-cells; Test type: Superiority or Other; p = 0.5595, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 7: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.3817, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 8: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.3623, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 9: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Double-negative B-cells; Test type: Superiority or Other; p = 0.7108, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 10: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Plasmablasts; Test type: Superiority or Other; p = 0.0639, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 11: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Naive B-cell compartment; Test type: Superiority or Other; p = 0.0186, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 12: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Transitional B-cells; Test type: Superiority or Other; p = 0.0050, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 13: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Naive B-cells; Test type: Superiority or Other; p = 0.0463, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 14: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Memory B-cells; Test type: Superiority or Other; p = 0.1919, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 15: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.3071, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 16: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Post-switch memory B-cells; Test type: Superiority or Other; p = 0.1714, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 17: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.1746, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 18: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.1626, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 19: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Double-negative B-cells; Test type: Superiority or Other; p = 0.6304, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 20: Comparison: TCZ/TCZ or TCZ/RTX; Week 24, Plasmablasts; Test type: Superiority or Other; p = 0.3449, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 21: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Naive B-cell compartment; Test type: Superiority or Other; p = 0.0919, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 22: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Transitional B-cells; Test type: Superiority or Other; p = 0.2189, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 23: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Naive B-cells; Test type: Superiority or Other; p = 0.1386, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 24: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Memory B-cells; Test type: Superiority or Other; p = 0.6199, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 25: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.1019, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 26: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Post-switch memory B-cells; Test type: Superiority or Other; p = 0.4353, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 27: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.3934, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 28: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.4196, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 29: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Double-negative B-cells; Test type: Superiority or Other; p = 0.5546, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 30: Comparison: TCZ/TCZ or TCZ/RTX; Week 32, Plasmablasts; Test type: Superiority or Other; p = 0.7695, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]

39. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Percentage of B-Cells at Baseline and Difference in DAS28 Scores Between Baseline and Weeks 16, 32, 40, 48, and 66 Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 38
Time Frame: Baseline and Weeks 16, 32, 40, 48, and 66
Population: ITT3 Population; n = number of data pairs included in the analysis.
Measure: Number; unit: coefficient
Units Other Than Participants: Pairs
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 27
Number analyzed (Pairs) | 24
coefficient
  Week 16, Naive B-cell compartment (n=24) | 0.09611
  Week 16, Transitional B-cells (n=24) | 0.08571
  Week 16, Naive B-cells (n=24) | 0.00870
  Week 16, Memory B-cells (n=6) | -0.60000
  Week 16, Pre-switch memory B-cells (n=24) | -0.15217
  Week 16, Post-switch memory B-cells (n=24) | -0.04004
  Week 16, IgG-positive class-switched (n=24) | -0.07528
  Week 16, IgA-positive class-switched (n=24) | 0.27049
  Week 16, Double-negative B-cells (n=6) | -0.14286
  Week 16, Plasmablasts (n=24) | 0.13232
  Week 32, Naive B-cell compartment (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Transitional B-cells (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Naive B-cells (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Memory B-cells (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Pre-switch memory B-cells (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Post-switch memory B-cells (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, IgG-positive class-switched (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, IgA-positive class-switched (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Double-negative B-cells (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 32, Plasmablasts (n=0) | NA — Participants in this population were followed for changes in DAS28 up to Week 16 compared to Baseline, and for changes up to Week 66 compared to Week 16. Thus, change from Baseline to Week 32 was not determined.
  Week 40, Naive B-cell compartment (n=2) | 1.00000
  Week 40, Transitional B-cells (n=2) | -1.00000
  Week 40, Naive B-cells (n=2) | 1.00000
  Week 40, Memory B-cells (n=0) | NA — Unable to calculate because the number of pairs was 0 at this assessment.
  Week 40, Pre-switch memory B-cells (n=2) | 1.00000
  Week 40, Post-switch memory B-cells (n=2) | 1.00000
  Week 40, IgG-positive class-switched (n=2) | 1.00000
  Week 40, IgA-positive class-switched (n=2) | 1.00000
  Week 40, Double-negative B-cells (n=0) | NA — Unable to calculate because the number of pairs was 0 at this assessment.
  Week 40, Plasmablasts (n=2) | 1.00000
  Week 48, Naive B-cell compartment (n=5) | 0.30000
  Week 48, Transitional B-cells (n=5) | -0.60000
  Week 48, Naive B-cells (n=5) | 0.30000
  Week 48, Memory B-cells (n=1) | NA — Unable to calculate because the number of pairs was 1 at this assessment.
  Week 48, Pre-switch memory B-cells (n=5) | 0.60000
  Week 48, Post-switch memory B-cells (n=5) | 0.20000
  Week 48, IgG-positive class-switched (n=5) | 0.20000
  Week 48, IgA-positive class-switched (n=5) | 0.50000
  Week 48, Double-negative B-cells (n=1) | NA — Unable to calculate because the number of pairs was 1 at this assessment.
  Week 48, Plasmablasts (n=5) | 0.10000
  Week 66, Naive B-cell compartment (n=10) | 0.12727
  Week 66, Transitional B-cells (n=10) | -0.03030
  Week 66, Naive B-cells (n=10) | 0.04242
  Week 66, Memory B-cells (n=3) | 1.00000
  Week 66, Pre-switch memory B-cells (n=10) | -0.03030
  Week 66, Post-switch memory B-cells (n=10) | 0.16364
  Week 66, IgG-positive class-switched (n=10) | 0.07295
  Week 66, IgA-positive class-switched (n=10) | 0.12805
  Week 66, Double-negative B-cells (n=3) | 1.00000
  Week 66, Plasmablasts (n=10) | 0.30909
Statistical Analysis 1: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Naive B-cell compartment; Test type: Superiority or Other; p = 0.6551, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 2: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Transitional B-cells; Test type: Superiority or Other; p = 0.6905, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Naive B-cells; Test type: Superiority or Other; p = 0.9678, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 4: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Memory B-cells; Test type: Superiority or Other; p = 0.2080, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 5: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.4778, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 6: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Post-switch memory B-cells; Test type: Superiority or Other; p = 0.8526, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 7: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.7266, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 8: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.2011, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 9: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Double-negative B-cells; Test type: Superiority or Other; p = 0.7872, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 10: Comparison: TCZ/TCZ or TCZ/RTX; Week 16, Plasmablasts; Test type: Superiority or Other; p = 0.5377, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 11: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, Naive B-cell compartment; Test type: Superiority or Other; p = 0.6238, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 12: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, Transitional B-cells; Test type: Superiority or Other; p = 0.2848, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 13: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, Naive B-cells; Test type: Superiority or Other; p = 0.6238, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 14: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.2848, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 15: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, Post-switch memory B-cells; Test type: Superiority or Other; p = 0.7471, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 16: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.7471, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 17: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.3910, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 18: Comparison: TCZ/TCZ or TCZ/RTX; Week 48, Plasmablasts; Test type: Superiority or Other; p = 0.8729, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 19: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Naive B-cell compartment; Test type: Superiority or Other; p = 0.7261, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 20: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Transitional B-cells; Test type: Superiority or Other; p = 0.9338, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 21: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Naive B-cells; Test type: Superiority or Other; p = 0.9074, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 22: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Memory B-cells; Test type: Superiority or Other; p < 0.0001, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 23: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Pre-switch memory B-cells; Test type: Superiority or Other; p = 0.9338, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 24: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Post-switch memory B-cells; Test type: Superiority or Other; p = 0.6515, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 25: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, IgG-positive class-switched B-cells; Test type: Superiority or Other; p = 0.8413, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 26: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, IgA-positive class-switched B-cells; Test type: Superiority or Other; p = 0.7244, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 27: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Double-negative B-cells; Test type: Superiority or Other; p < 0.0001, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]
Statistical Analysis 28: Comparison: TCZ/TCZ or TCZ/RTX; Week 66, Plasmablasts; Test type: Superiority or Other; p = 0.3848, Spearman Rank-Order Correlation; [statistical method as in outcome 37, analysis 1]

40. Secondary Outcome: Mean Number of Work Days Missed Per Week
Description: Work days missed were documented by reason (either rheumatoid arthritis [RA] or other reasons) for each participant over the preceding 7-day period. The mean number of work days missed was calculated by averaging the number of days missed per week among all participants.
Time Frame: Baseline and Week 16
Population: Main ITT Population. Employed participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 241
days
  Due to RA, Baseline (n=241) | 1.03 (2.30)
  Due to RA, Week 16 (n=221) | 0.39 (1.51)
  Due to other reasons, Baseline (n=233) | 0.14 (0.87)
  Due to other reasons, Week 16 (n=222) | 0.32 (1.26)

41. Secondary Outcome: Quality of Life as Assessed Using Short Form 36 (SF-36)
Description: The SF-36 evaluates participant-rated quality of life using 8 domains: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for each section is the average of the individual question scores, which are scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants.
Time Frame: Baseline and Week 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 513
units on a scale
  Physical functioning, Baseline (n=511) | 49.6 (23.7)
  Physical functioning, Week 16 (n=473) | 64.1 (25.5)
  Role (physical), Baseline (n=508) | 12.9 (18.1)
  Role (physical), Week 16 (n=472) | 29.9 (21.4)
  Bodily pain, Baseline (n=512) | 31.3 (18.2)
  Bodily pain, Week 16 (n=474) | 55.3 (17.8)
  General health, Baseline (n=504) | 43.6 (16.7)
  General health, Week 16 (n=468) | 54.3 (18.3)
  Vitality, Baseline (n=512) | 44.0 (19.7)
  Vitality, Week 16 (n=474) | 58.1 (20.4)
  Social functioning, Baseline (n=507) | 68.1 (24.8)
  Social functioning, Week 16 (n=464) | 80.1 (21.6)
  Role (emotional), Baseline (n=505) | 55.9 (45.0)
  Role (emotional), Week 16 (n=472) | 70.9 (42.1)
  Mental health, Baseline (n=513) | 63.5 (18.7)
  Mental health, Week 16 (n=474) | 72.3 (17.9)

42. Secondary Outcome: Change From Baseline in Quality of Life as Assessed Using SF-36 at Week 16
Description: The SF-36 evaluates participant-rated quality of life using 8 domains: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for each section is the average of the individual question scores, which are scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants, and the change in each domain score was calculated as [mean score at Week 16 minus mean score at Baseline].
Time Frame: Baseline and Week 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 470
units on a scale
  Physical functioning (n=466) | 14.3 (21.8)
  Role (physical) (n=461) | 17.0 (22.0)
  Bodily pain (n=470) | 23.9 (21.1)
  General health (n=454) | 10.4 (18.5)
  Vitality (n=468) | 13.9 (19.3)
  Social functioning (n=456) | 12.0 (23.8)
  Role (emotional) (n=459) | 14.7 (46.1)
  Mental health (n=468) | 8.7 (16.8)

43. Secondary Outcome: Change From Week 16 to 32 in Quality of Life as Assessed Using SF-36 Scores Among Participants Treated With 8 Courses of Tocilizumab
Description: The SF-36 evaluates participant-rated quality of life using 8 domains: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for each section is the average of the individual question scores, which are scaled from 0 to 100, with higher scores indicating better functioning. The mean score at each timepoint was determined by averaging the scores among all participants, and the change in each domain score was calculated as [mean score at Week 32 minus mean score at Week 16].
Time Frame: Weeks 16 and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 188
units on a scale
  Physical functioning (n=188) | 3.6 (16.6)
  Role (physical) (n=187) | 2.0 (20.6)
  Bodily pain (n=188) | 3.2 (16.5)
  General health (n=184) | 2.6 (14.3)
  Vitality (n=186) | 2.7 (14.2)
  Social functioning (n=184) | -0.3 (19.6)
  Role (emotional) (n=184) | 5.5 (42.3)
  Mental health (n=186) | 0.7 (15.3)

44. Secondary Outcome: Change From Week 16 to 32 in Quality of Life as Assessed Using SF-36 Scores Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 43
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 26
units on a scale
  Physical functioning (n=26) | 2.5 (20.0)
  Role (physical) (n=24) | -1.0 (21.5)
  Bodily pain (n=26) | 10.6 (20.8)
  General health (n=24) | 5.2 (18.1)
  Vitality (n=26) | 1.0 (9.3)
  Social functioning (n=24) | -3.1 (17.4)
  Role (emotional) (n=24) | 2.8 (35.3)
  Mental health (n=26) | 3.4 (10.7)

45. Secondary Outcome: Quality of Life as Assessed Using HAQ-DI
Description: The HAQ-DI evaluates participant-reported quality of life using 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities such as running errands and performing household chores. Each category contains multiple questions, which are answered using a 4-point scale from 0 to 3. The overall index score is taken as an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. The mean index score at each timepoint was determined by averaging the scores among all participants.
Time Frame: Baseline and Week 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 513
units on a scale
  Baseline (n=513) | 1.24 (0.67)
  Week 16 (n=472) | 0.75 (0.67)

46. Secondary Outcome: Change From Baseline in Quality of Life as Assessed Using HAQ-DI at Week 16
Description: The HAQ-DI evaluates participant-reported quality of life using 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities such as running errands and performing household chores. Each category contains multiple questions, which are answered using a 4-point scale from 0 to 3. The overall index score is taken as an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. The mean index score at each timepoint was determined by averaging the scores among all participants, and the change in score was calculated as [mean score at Week 16 minus mean score at Baseline].
Time Frame: Baseline and Week 16
Population: Main ITT Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 466
units on a scale | -0.48 (0.58)

47. Secondary Outcome: Change From Week 16 to 32 in Quality of Life as Assessed Using HAQ-DI Among Participants Treated With 8 Courses of Tocilizumab
Description: The HAQ-DI evaluates participant-reported quality of life using 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities such as running errands and performing household chores. Each category contains multiple questions, which are answered using a 4-point scale from 0 to 3. The overall index score is taken as an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. The mean index score at each timepoint was determined by averaging the scores among all participants, and the change in score was calculated as [mean score at Week 32 minus the mean score at Week 16].
Time Frame: Weeks 16 and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 187
units on a scale | -0.06 (0.34)

48. Secondary Outcome: Change From Week 16 to 32 in Quality of Life as Assessed Using HAQ-DI Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 47
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 26
units on a scale | -0.10 (0.39)

49. Secondary Outcome: Percentage of Participants Achieving a Response According to HAQ-DI Criteria
Description: The HAQ-DI evaluates participant-reported quality of life using 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities such as running errands and performing household chores. Each category contains multiple questions, which are answered using a 4-point scale from 0 to 3. The overall index score is taken as an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. Response was defined as a change in index score >0.22 from Baseline to Week 16.
Time Frame: Baseline and Week 16
Population: Main ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 519
percentage of participants | 61.1

50. Secondary Outcome: Quality of Life as Assessed Using Functional Assessment of Chronic Illness Therapy (FACIT)
Description: The FACIT-F evaluates quality of life using 5 categories: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and fatigue (FS). Participants answer each item on a 5-point scale from 0 to 4. The total score is the sum of individual responses across all 5 categories and may range from 0 to 160. The FACIT-General (FACIT-G; range 0 to 108) is the sum of scores for PWB, SWB, EWB, and FWB; the FACIT-Fatigue (FACIT-F) trial outcome index (TOI; range 0 to 108) is the sum of scores for PWB, FWB, and FS; and the FACIT-F fatigue (range 0 to 52) is the sum of scores for the FS only. For derivations of the FACIT-F reported here, higher scores indicate better quality of life. The mean score at each timepoint was determined by averaging scores among all participants.
Time Frame: Baseline and Week 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 510
units on a scale
  FACIT-F TOI, Baseline (n=498) | 66.2 (20.6)
  FACIT-F TOI, Week 16 (n=460) | 80.8 (19.3)
  FACIT-G total, Baseline (n=498) | 71.1 (15.7)
  FACIT-G total, Week 16 (n=462) | 82.6 (15.9)
  FACIT-F total, Baseline (n=494) | 103.8 (25.5)
  FACIT-F total, Week 16 (n=458) | 121.9 (25.3)
  FACIT-F fatigue, Baseline (n=510) | 32.7 (11.6)
  FACIT-F fatigue, Week 16 (n=475) | 39.2 (10.6)

51. Secondary Outcome: Change From Baseline in Quality of Life as Assessed Using FACIT at Week 16
Description: The FACIT-F evaluates quality of life using 5 categories: PWB, SWB, EWB, FWB, and FS. Participants answer each item on a 5-point scale from 0 to 4. The total score is the sum of individual responses across all 5 categories and may range from 0 to 160. The FACIT-G (range 0 to 108) is the sum of scores for PWB, SWB, EWB, and FWB; the FACIT-F TOI (range 0 to 108) is the sum of scores for PWB, FWB, and FS; and the FACIT-F fatigue (range 0 to 52) is the sum of scores for the FS only. For derivations of the FACIT-F reported here, higher scores indicate better quality of life. The mean score at each timepoint was determined by averaging scores among all participants, and the change in score was calculated as [mean score at Week 16 minus mean score at Baseline].
Time Frame: Baseline and Week 16
Population: Main ITT Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 467
units on a scale
  FACIT-F TOI (n=445) | 14.2 (17.9)
  FACIT-G total (n=445) | 10.8 (13.6)
  FACIT-F total (n=439) | 17.5 (21.8)
  FACIT-F fatigue (n=467) | 6.6 (9.9)

52. Secondary Outcome: Change From Week 16 to 32 in Quality of Life as Assessed Using FACIT Among Participants Treated With 8 Courses of Tocilizumab
Description: The FACIT-F evaluates quality of life using 5 categories: PWB, SWB, EWB, FWB, and FS. Participants answer each item on a 5-point scale from 0 to 4. The total score is the sum of individual responses across all 5 categories and may range from 0 to 160. The FACIT-G (range 0 to 108) is the sum of scores for PWB, SWB, EWB, and FWB; the FACIT-F TOI (range 0 to 108) is the sum of scores for PWB, FWB, and FS; and the FACIT-F fatigue (range 0 to 52) is the sum of scores for the FS only. For derivations of the FACIT-F reported here, higher scores indicate better quality of life. The mean score at each timepoint was determined by averaging scores among all participants, and the change in score was calculated as [mean score at Week 32 minus mean score at Week 16].
Time Frame: Weeks 16 and 32
Population: ITT2 Population. Participants with evaluable data at the designated visit (number shown = n) were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 186
units on a scale
  FACIT-F TOI (n=172) | 1.7 (12.9)
  FACIT-G total (n=174) | 1.1 (9.2)
  FACIT-F total (n=170) | 2.0 (15.1)
  FACIT-F fatigue (n=186) | 0.8 (7.4)

53. Secondary Outcome: Change From Week 16 to 32 in Quality of Life as Assessed Using FACIT Among Nonresponding Participants Treated With Rituximab
Description: as for outcome 52
Time Frame: Weeks 16 and 32
Population: ITT3 Population. Participants with evaluable data at the designated visit were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ/TCZ or TCZ/RTX
Number analyzed (Participants) | 26
units on a scale
  FACIT-F TOI | 2.9 (9.8)
  FACIT-G total | 3.0 (8.3)
  FACIT-F total | 4.4 (12.5)
  FACIT-F fatigue | 1.4 (5.8)

ADVERSE EVENTS:
Time Frame: Up to 66 weeks
Description: Adverse events (AEs) were assessed at each treatment visit from Baseline to Week 16, at which point participants having achieved early remission completed the study. Those who did not achieve early remission continued to receive treatment, and AEs were assessed until 4 weeks after last dose (TCZ/TCZ) or until Week 66 (TCZ/RTX).
Arm/Group | TCZ/TCZ or TCZ/RTX
Serious Adverse Events (participants affected / at risk) | 54/519
Other Adverse Events (participants affected / at risk) | 104/519
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ/TCZ or TCZ/RTX (N=519)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Fibrin D dimer increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Intracranial haematoma (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ/TCZ or TCZ/RTX (N=519)
Nasopharyngitis (Infections and infestations) | 77
Hypertension (Vascular disorders) | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.